CLINICAL TRIAL: NCT06289218
Title: Kinesio Taping Versus Interferential Current Therapy in Treating Knee Osteoarthritis: a Comparative Study
Brief Title: Kinesio Taping Versus Interferential Current Therapy in Treating Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Norhan Elsaid Ahmed Elsaid, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Treating knee osteoarthritis
Record Dates: First submitted 2024-02-18; First posted 2024-03-01 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Electric Stimulation Therapy; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- interferential current plus exercise (Experimental): interferential current plus exercise group
  Interventions: Device: interferential current
- kinesio taping plus exercise (Experimental): kinesio taping plus exercise group
  Interventions: Other: kinesio taping
- Control group (Other): Control group
  Interventions: Other: exercise

INTERVENTIONS:
Device: interferential current — IFC plus exercise
  Other Names: IFC
  Arms: interferential current plus exercise
Other: kinesio taping — KT plus exercise
  Other Names: KT
  Arms: kinesio taping plus exercise
Other: exercise — exercise only
  Arms: Control group

SUMMARY:
The purpose of this study will be to compare the combined effect of using Kinesio taping versus interferential current with an exercise program on knee pain, function, knee range of motion, knee muscle strength, and functional mobility in chronic knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is the most common form of degenerative joint disease affecting 15%-40% of people over 40 years of age. In 2020, the global incidence of KOA was 86.7 million individuals. KOA is responsible for substantial health and economic costs. KOA is the most common cause of pain and disability among older persons. The key symptoms of KOA are pain, functional disability, and decreased patient quality of life through its negative effects on mobility, mood, and sleep. Other symptoms are swelling, stiffness, joint deformity, and muscular atrophy.

The Treatment goals for KOA are to decrease pain and improve physical function. Physical therapy decreased pain and functional disability in patients with KOA. The therapeutic techniques include therapeutic exercises, electrotherapy, and manual therapy. Several meta-analysis and systematic reviews have evidence of various types of exercises including aerobic and resistance exercises which is effective in reducing pain and functional disabilities in a patient with KOA especially quadriceps muscle strengthening with open and closed chain training. Specific recommendations including physical activity, reducing body weight, reducing sedentary time, and managing diabetes disease can improve function and symptoms of KOA. To improve the individual's function, and reduce pain and disability, several interventions had been investigated to promote physical activity.

Kinesio taping (KT) is a conservative therapeutic technique used for the treatment of several musculoskeletal disorders which has increased attention from physicians and physiotherapists in recent years. KT, first introduced in 1979 in Japan, is used for the treatment and prevention of several sports injuries and several clinical conditions. In 2011, KT is recommended by the American College of Rheumatology (ACR) for the treatment of patients with knee OA, and it is commonly used to treat knee OA.

Kinesio taping (KT) is an alternative taping technique which is an elastic woven cotton strip with heat-sensitive acrylic adhesive, a high-stretch elastic adhesive material, it is applied directly to the skin and can be left on the skin for several days due to its strong adherence. The application of KT for four weeks can reduce the pain so the patient can reduce the use pain killers. Kinesio taping (KT) is a low-cost, safe, noninvasive, non-pharmacological method, that has minimal side effects and can be a convenient option for the treatment of musculoskeletal disorders such as knee OA.

Interferential current (IFC) is a simple, non-invasive, non-pharmacological, more comfortable treatment used to relieve pain. IFC known as kilohertz-frequency alternating current, which is a pair of signal generators with one fixed frequency of 4000 Hz and the other varying in frequency between 4000 and 4250 Hz. IFC can reduce skin impedance, reach deeper tissue, and can be utilized as an alternative medication or supplement to drugs in treating pain. IFC is the most effective pain relief treatment for the management of KOA.

Exercises play a major role in treating patients with KOA; it can improve both pain and function. Therefore What about comparing the application of kinesio taping combined with exercises versus the IFC therapy combined with exercises in treating patients with KOA?

ELIGIBILITY:
Inclusion Criteria:

* sixty-three Male and female patients aged between 40 and 65 years old were diagnosed clinically and radiologically as knee osteoarthritis grade mild and moderate chronic knee osteoarthritis.
* BMI ranges between 20 and 32 kg/m2.
* Knee OA grades 1 and 2 are based on Kellgren and Lawrence's grades. Narrowing of joint space, definite osteophytes.
* Unilateral knee osteoarthritis.
* Knee pain for most days of the prior month, in addition to at least 3 of the following:

  1. Crepitus on active joint motion
  2. Morning stiffness less than 30 minutes duration
  3. Age older than 50 years
  4. Bony enlargement of the knee on examination
  5. Bony tenderness of the knee on examination
  6. No palpable warmth.

Exclusion Criteria:

* Patients having the following conditions will be excluded from the study:

  * Comorbidities such as (rheumatoid arthritis, cancer, osteoporosis, and joint infection).
  * Previous surgery for knee OA.
  * BMI more than 33 kg/m2.
  * Suffering from polyarticular disease.
  * Severe mechanical deformity (diaphyseal Varus deformity of 4° and valgus of 16°).
  * Previous arthroscopy within the last year.
  * Systemic autoimmune rheumatoid disease (connective tissue disease and systemic necrotizing vasculitis).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-09-21 (Estimated); Study Completion 2025-09-21 (Estimated)

PRIMARY OUTCOMES:
knee flexion range of motion | pre-intervention and after 4 weeks of treatment
  to measure Knee joint active range of motion (flexion) by universal goniometer
knee extension range of motion | pre-intervention and after 4 weeks of treatment
  to measure Knee joint active range of motion (extension) by universal goniometer
quadriceps muscle strength | pre-intervention and after 4 weeks of treatment
  to test the isometric quadriceps muscle strength by hand-held dynamometer
The Western Ontario and McMaster Universities Osteoarthritis Index | pre-intervention and after 4 weeks of treatment
  to measure knee function and knee pain degree
Timed up and go test | pre-intervention and after 4 weeks of treatment
  to measure knee function mobility by the Timed up and go test

CONTACTS AND LOCATIONS:
Overall Officials: Salwa Fadl Abd Elmageed, Prof.Dr, Principal Investigator — Professor at Department of Physical Therapy for Musculoskeletal Disorders and Its Surgery

REFERENCES:
- [Background] Aaron RK, Ciombor DM. Therapeutic effects of electromagnetic fields in the stimulation of connective tissue repair. J Cell Biochem. 1993 May;52(1):42-6. doi: 10.1002/jcb.240520107. PMID 8320274
- [Background] Alqualo-Costa R, Thome GR, Perracini MR, Liebano RE. Low-level laser therapy and interferential current in patients with knee osteoarthritis: a randomized controlled trial protocol. Pain Manag. 2018 May;8(3):157-166. doi: 10.2217/pmt-2017-0057. Epub 2018 May 3. PMID 29722602
- [Background] Atamaz FC, Durmaz B, Baydar M, Demircioglu OY, Iyiyapici A, Kuran B, Oncel S, Sendur OF. Comparison of the efficacy of transcutaneous electrical nerve stimulation, interferential currents, and shortwave diathermy in knee osteoarthritis: a double-blind, randomized, controlled, multicenter study. Arch Phys Med Rehabil. 2012 May;93(5):748-56. doi: 10.1016/j.apmr.2011.11.037. Epub 2012 Mar 28. PMID 22459699
- [Background] Aw NM, Yeo SJ, Wylde V, Wong SB, Chan D, Thumboo J, Leung YY. Impact of pain sensitisation on the quality of life of patients with knee osteoarthritis. RMD Open. 2022 Mar;8(1):e001938. doi: 10.1136/rmdopen-2021-001938. PMID 35296529
- [Background] Beauchet O, Fantino B, Allali G, Muir SW, Montero-Odasso M, Annweiler C. Timed Up and Go test and risk of falls in older adults: a systematic review. J Nutr Health Aging. 2011 Dec;15(10):933-8. doi: 10.1007/s12603-011-0062-0. PMID 22159785
- [Background] Brunenberg DE, van Steyn MJ, Sluimer JC, Bekebrede LL, Bulstra SK, Joore MA. Joint recovery programme versus usual care: an economic evaluation of a clinical pathway for joint replacement surgery. Med Care. 2005 Oct;43(10):1018-26. doi: 10.1097/01.mlr.0000178266.75744.35. PMID 16166871
- [Background] Cadogan A, Laslett M, Hing W, McNair P, Williams M. Reliability of a new hand-held dynamometer in measuring shoulder range of motion and strength. Man Ther. 2011 Feb;16(1):97-101. doi: 10.1016/j.math.2010.05.005. PMID 20621547
- [Background] Celik D, Dirican A, Baltaci G. Intrarater reliability of assessing strength of the shoulder and scapular muscles. J Sport Rehabil. 2012 Feb 29;21(1):1-5. doi: 10.1123/jsr.2012.TR3. Print 2012 Feb 1. PMID 22495260
- [Background] Chapple CM, Nicholson H, Baxter GD, Abbott JH. Patient characteristics that predict progression of knee osteoarthritis: a systematic review of prognostic studies. Arthritis Care Res (Hoboken). 2011 Aug;63(8):1115-25. doi: 10.1002/acr.20492. PMID 21560257
- [Background] Chen HL, Yang FA, Lee TH, Liou TH, Escorpizo R, Chen HC. Effectiveness of interferential current therapy in patients with knee osteoarthritis: a systematic review and meta-analysis of randomized controlled trials. Sci Rep. 2022 Jun 11;12(1):9694. doi: 10.1038/s41598-022-13478-6. PMID 35690604
- [Background] de Paula Gomes CAF, Politti F, de Souza Bacelar Pereira C, da Silva ACB, Dibai-Filho AV, de Oliveira AR, Biasotto-Gonzalez DA. Exercise program combined with electrophysical modalities in subjects with knee osteoarthritis: a randomised, placebo-controlled clinical trial. BMC Musculoskelet Disord. 2020 Apr 20;21(1):258. doi: 10.1186/s12891-020-03293-3. PMID 32312265
- [Background] Deyle GD, Allen CS, Allison SC, Gill NW, Hando BR, Petersen EJ, Dusenberry DI, Rhon DI. Physical Therapy versus Glucocorticoid Injection for Osteoarthritis of the Knee. N Engl J Med. 2020 Apr 9;382(15):1420-1429. doi: 10.1056/NEJMoa1905877. PMID 32268027
- [Background] Ellison AE, Berg EE. Embryology, anatomy, and function of the anterior cruciate ligament. Orthop Clin North Am. 1985 Jan;16(1):3-14. PMID 3969275
- [Background] Escamilla RF, Zheng N, Macleod TD, Edwards WB, Hreljac A, Fleisig GS, Wilk KE, Moorman CT 3rd, Imamura R, Andrews JR. Patellofemoral joint force and stress between a short- and long-step forward lunge. J Orthop Sports Phys Ther. 2008 Nov;38(11):681-90. doi: 10.2519/jospt.2008.2694. PMID 18978453
- [Background] Goats GC. Pulsed electromagnetic (short-wave) energy therapy. Br J Sports Med. 1989 Dec;23(4):213-6. doi: 10.1136/bjsm.23.4.213. No abstract available. PMID 2629997
- [Background] Goats GC. Interferential current therapy. Br J Sports Med. 1990 Jun;24(2):87-92. doi: 10.1136/bjsm.24.2.87. No abstract available. PMID 1702337
- [Background] Goldring MB, Goldring SR. Articular cartilage and subchondral bone in the pathogenesis of osteoarthritis. Ann N Y Acad Sci. 2010 Mar;1192:230-7. doi: 10.1111/j.1749-6632.2009.05240.x. PMID 20392241
- [Background] Goldring MB, Marcu KB. Cartilage homeostasis in health and rheumatic diseases. Arthritis Res Ther. 2009;11(3):224. doi: 10.1186/ar2592. Epub 2009 May 19. PMID 19519926
- [Background] Goldring SR, Goldring MB. Changes in the osteochondral unit during osteoarthritis: structure, function and cartilage-bone crosstalk. Nat Rev Rheumatol. 2016 Nov;12(11):632-644. doi: 10.1038/nrrheum.2016.148. Epub 2016 Sep 22. PMID 27652499
- [Background] Gruber J, Wolter D, Lierse W. [Anterior cruciate ligament reflex (LCA reflex)]. Unfallchirurg. 1986 Dec;89(12):551-4. No abstract available. German. PMID 3563529
- [Background] Guermazi M, Poiraudeau S, Yahia M, Mezganni M, Fermanian J, Habib Elleuch M, Revel M. Translation, adaptation and validation of the Western Ontario and McMaster Universities osteoarthritis index (WOMAC) for an Arab population: the Sfax modified WOMAC. Osteoarthritis Cartilage. 2004 Jun;12(6):459-68. doi: 10.1016/j.joca.2004.02.006. PMID 15135142
- [Background] Gunaydin OE, Bayrakci Tunay V. Comparison of the added effects of kinesio taping and extracorporeal shockwave therapy to exercise alone in knee osteoarthritis. Physiother Theory Pract. 2022 May;38(5):661-669. doi: 10.1080/09593985.2020.1780657. Epub 2020 Jun 23. PMID 32574094
- [Background] Gundog M, Atamaz F, Kanyilmaz S, Kirazli Y, Celepoglu G. Interferential current therapy in patients with knee osteoarthritis: comparison of the effectiveness of different amplitude-modulated frequencies. Am J Phys Med Rehabil. 2012 Feb;91(2):107-13. doi: 10.1097/PHM.0b013e3182328687. PMID 22019968
- [Background] Hamilton DF, Akhtar S, Griffiths B, Prior Y, Jones RK. The use of technology to support lifestyle interventions in knee osteoarthritis: A scoping review. Osteoarthr Cartil Open. 2023 Feb 9;5(2):100344. doi: 10.1016/j.ocarto.2023.100344. eCollection 2023 Jun. PMID 36852286
- [Background] Hancock GE, Hepworth T, Wembridge K. Accuracy and reliability of knee goniometry methods. J Exp Orthop. 2018 Oct 19;5(1):46. doi: 10.1186/s40634-018-0161-5. PMID 30341552
- [Background] Hirano M, Katoh M, Gomi M, Arai S. Validity and reliability of isometric knee extension muscle strength measurements using a belt-stabilized hand-held dynamometer: a comparison with the measurement using an isokinetic dynamometer in a sitting posture. J Phys Ther Sci. 2020 Feb;32(2):120-124. doi: 10.1589/jpts.32.120. Epub 2020 Feb 14. PMID 32158074
- [Background] Hirschmann MT, Muller W. Complex function of the knee joint: the current understanding of the knee. Knee Surg Sports Traumatol Arthrosc. 2015 Oct;23(10):2780-8. doi: 10.1007/s00167-015-3619-3. Epub 2015 May 12. PMID 25962963
- [Background] Johansson H, Sjolander P, Sojka P. A sensory role for the cruciate ligaments. Clin Orthop Relat Res. 1991 Jul;(268):161-78. PMID 2060205
- [Background] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- [Background] Lee R, Kean WF. Obesity and knee osteoarthritis. Inflammopharmacology. 2012 Apr;20(2):53-8. doi: 10.1007/s10787-011-0118-0. Epub 2012 Jan 12. PMID 22237485
- [Background] Lehman GJ, Hoda W, Oliver S. Trunk muscle activity during bridging exercises on and off a Swiss ball. Chiropr Osteopat. 2005 Jul 30;13:14. doi: 10.1186/1746-1340-13-14. PMID 16053529
- [Background] Lenssen AF, van Dam EM, Crijns YH, Verhey M, Geesink RJ, van den Brandt PA, de Bie RA. Reproducibility of goniometric measurement of the knee in the in-hospital phase following total knee arthroplasty. BMC Musculoskelet Disord. 2007 Aug 17;8:83. doi: 10.1186/1471-2474-8-83. PMID 17705860
- [Background] Lespasio MJ, Piuzzi NS, Husni ME, Muschler GF, Guarino A, Mont MA. Knee Osteoarthritis: A Primer. Perm J. 2017;21:16-183. doi: 10.7812/TPP/16-183. PMID 29035179
- [Background] Lin CH, Lee M, Lu KY, Chang CH, Huang SS, Chen CM. Comparative effects of combined physical therapy with Kinesio taping and physical therapy in patients with knee osteoarthritis: a systematic review and meta-analysis. Clin Rehabil. 2020 Aug;34(8):1014-1027. doi: 10.1177/0269215520928398. Epub 2020 Jun 28. PMID 32597199
- [Background] Lu Z, Li X, Chen R, Guo C. Kinesio taping improves pain and function in patients with knee osteoarthritis: A meta-analysis of randomized controlled trials. Int J Surg. 2018 Nov;59:27-35. doi: 10.1016/j.ijsu.2018.09.015. Epub 2018 Sep 28. PMID 30273684
- [Background] Mansfield JC, Winlove CP. A multi-modal multiphoton investigation of microstructure in the deep zone and calcified cartilage. J Anat. 2012 Apr;220(4):405-16. doi: 10.1111/j.1469-7580.2012.01479.x. Epub 2012 Feb 14. PMID 22332832
- [Background] Mao HY, Hu MT, Yen YY, Lan SJ, Lee SD. Kinesio Taping Relieves Pain and Improves Isokinetic Not Isometric Muscle Strength in Patients with Knee Osteoarthritis-A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Oct 4;18(19):10440. doi: 10.3390/ijerph181910440. PMID 34639740
- [Background] McCloskey DI, Cross MJ, Honner R, Potter EK. Sensory effects of pulling or vibrating exposed tendons in man. Brain. 1983 Mar;106 (Pt 1):21-37. doi: 10.1093/brain/106.1.21. PMID 6831197
- [Background] McConnell S, Kolopack P, Davis AM. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): a review of its utility and measurement properties. Arthritis Rheum. 2001 Oct;45(5):453-61. doi: 10.1002/1529-0131(200110)45:53.0.co;2-w. No abstract available. PMID 11642645
- [Background] Mitra, M., & Gaikwad, N. (2019). The Effect of Straight Leg Raise with Lumbar Stabilization Exercises in Subjects of Low Back Pain with Adverse Neural Tension between the Age Group 20-50 Years. Executive Editor, 13(1), 101.
- [Background] Mohamed SHP, Alatawi SF. Effectiveness of Kinesio taping and conventional physical therapy in the management of knee osteoarthritis: a randomized clinical trial. Ir J Med Sci. 2023 Oct;192(5):2223-2233. doi: 10.1007/s11845-022-03247-9. Epub 2022 Dec 17. PMID 36527538
- [Background] Morris S, Morris ME, Iansek R. Reliability of measurements obtained with the Timed "Up & Go" test in people with Parkinson disease. Phys Ther. 2001 Feb;81(2):810-8. doi: 10.1093/ptj/81.2.810. PMID 11175678
- [Background] Musumeci, G. (2016). The effect of mechanical loading on articular cartilage. Journal of Functional Morphology and Kinesiology, 1(2), 154-161.
- [Background] Kaya Mutlu E, Mustafaoglu R, Birinci T, Razak Ozdincler A. Does Kinesio Taping of the Knee Improve Pain and Functionality in Patients with Knee Osteoarthritis?: A Randomized Controlled Clinical Trial. Am J Phys Med Rehabil. 2017 Jan;96(1):25-33. doi: 10.1097/PHM.0000000000000520. PMID 27149590
- [Background] Parreira Pdo C, Costa Lda C, Hespanhol LC Jr, Lopes AD, Costa LO. Current evidence does not support the use of Kinesio Taping in clinical practice: a systematic review. J Physiother. 2014 Mar;60(1):31-9. doi: 10.1016/j.jphys.2013.12.008. Epub 2014 Apr 24. PMID 24856938
- [Background] Paul-Dauphin A, Guillemin F, Virion JM, Briancon S. Bias and precision in visual analogue scales: a randomized controlled trial. Am J Epidemiol. 1999 Nov 15;150(10):1117-27. doi: 10.1093/oxfordjournals.aje.a009937. PMID 10568628
- [Background] Pinto-Ramos J, Moreira T, Costa F, Tavares H, Cabral J, Costa-Santos C, Barroso J, Sousa-Pinto B. Handheld dynamometer reliability to measure knee extension strength in rehabilitation patients-A cross-sectional study. PLoS One. 2022 May 17;17(5):e0268254. doi: 10.1371/journal.pone.0268254. eCollection 2022. PMID 35580110
- [Background] Prathap Kumar, J., Arun Kumar, M., & Venkatesh, D. (2020). Healthy gait: Review of anatomy and physiology of knee joint. International Journal of Current Research and Review, 12(6), 1-8.
- [Background] Prentice AM, Jebb SA. Beyond body mass index. Obes Rev. 2001 Aug;2(3):141-7. doi: 10.1046/j.1467-789x.2001.00031.x. PMID 12120099
- [Background] Primorac D, Molnar V, Rod E, Jelec Z, Cukelj F, Matisic V, Vrdoljak T, Hudetz D, Hajsok H, Boric I. Knee Osteoarthritis: A Review of Pathogenesis and State-Of-The-Art Non-Operative Therapeutic Considerations. Genes (Basel). 2020 Jul 26;11(8):854. doi: 10.3390/genes11080854. PMID 32722615
- [Background] Rampazo EP, Liebano RE. Analgesic Effects of Interferential Current Therapy: A Narrative Review. Medicina (Kaunas). 2022 Jan 17;58(1):141. doi: 10.3390/medicina58010141. PMID 35056448
- [Background] Raposo F, Ramos M, Lucia Cruz A. Effects of exercise on knee osteoarthritis: A systematic review. Musculoskeletal Care. 2021 Dec;19(4):399-435. doi: 10.1002/msc.1538. Epub 2021 Mar 5. PMID 33666347
- [Background] Reginster, J. Y., Pelletier, J. P., Martel-Pelletier, J., Henrotin, Y., Crasborn, L., Crielaard, J. M., & Henrotin, Y. (1999). Scientific basis of physical therapy and rehabilitation in the management of patients with osteoarthritis. Osteoarthritis: Clinical and Experimental Aspects, 453-479.
- [Background] Rogind H, Bibow-Nielsen B, Jensen B, Moller HC, Frimodt-Moller H, Bliddal H. The effects of a physical training program on patients with osteoarthritis of the knees. Arch Phys Med Rehabil. 1998 Nov;79(11):1421-7. doi: 10.1016/s0003-9993(98)90238-6. PMID 9821904
- [Background] Ruhlen R, Marberry K. The chondrocyte primary cilium. Osteoarthritis Cartilage. 2014 Aug;22(8):1071-6. doi: 10.1016/j.joca.2014.05.011. Epub 2014 May 29. PMID 24879961
- [Background] Sanchez M, Fiz N, Azofra J, Usabiaga J, Aduriz Recalde E, Garcia Gutierrez A, Albillos J, Garate R, Aguirre JJ, Padilla S, Orive G, Anitua E. A randomized clinical trial evaluating plasma rich in growth factors (PRGF-Endoret) versus hyaluronic acid in the short-term treatment of symptomatic knee osteoarthritis. Arthroscopy. 2012 Aug;28(8):1070-8. doi: 10.1016/j.arthro.2012.05.011. PMID 22840987
- [Background] Shamsi M, Mirzaei M, Khabiri SS. Universal goniometer and electro-goniometer intra-examiner reliability in measuring the knee range of motion during active knee extension test in patients with chronic low back pain with short hamstring muscle. BMC Sports Sci Med Rehabil. 2019 Mar 22;11:4. doi: 10.1186/s13102-019-0116-x. eCollection 2019. PMID 30949343
- [Background] Suzuki K, Akasaka K, Otsudo T, Sawada Y, Hattori H, Hasebe Y, Mizoguchi Y, Hall TM, Yamamoto M. Effects of functional movement screen training in high-school baseball players: A randomized controlled clinical trial. Medicine (Baltimore). 2021 Apr 9;100(14):e25423. doi: 10.1097/MD.0000000000025423. PMID 33832142
- [Background] Tsokanos A, Livieratou E, Billis E, Tsekoura M, Tatsios P, Tsepis E, Fousekis K. The Efficacy of Manual Therapy in Patients with Knee Osteoarthritis: A Systematic Review. Medicina (Kaunas). 2021 Jul 7;57(7):696. doi: 10.3390/medicina57070696. PMID 34356977
- [Background] Tsuda E, Okamura Y, Otsuka H, Komatsu T, Tokuya S. Direct evidence of the anterior cruciate ligament-hamstring reflex arc in humans. Am J Sports Med. 2001 Jan-Feb;29(1):83-7. doi: 10.1177/03635465010290011801. PMID 11206261
- [Background] Turner MN, Hernandez DO, Cade W, Emerson CP, Reynolds JM, Best TM. The Role of Resistance Training Dosing on Pain and Physical Function in Individuals With Knee Osteoarthritis: A Systematic Review. Sports Health. 2020 Mar/Apr;12(2):200-206. doi: 10.1177/1941738119887183. Epub 2019 Dec 18. PMID 31850826
- [Background] Watkins MA, Riddle DL, Lamb RL, Personius WJ. Reliability of goniometric measurements and visual estimates of knee range of motion obtained in a clinical setting. Phys Ther. 1991 Feb;71(2):90-6; discussion 96-7. doi: 10.1093/ptj/71.2.90. PMID 1989012
- [Background] Wikholm JB, Bohannon RW. Hand-held Dynamometer Measurements: Tester Strength Makes a Difference. J Orthop Sports Phys Ther. 1991;13(4):191-8. doi: 10.2519/jospt.1991.13.4.191. PMID 18796845
- [Background] Wodowski AJ, Swigler CW, Liu H, Nord KM, Toy PC, Mihalko WM. Proprioception and Knee Arthroplasty: A Literature Review. Orthop Clin North Am. 2016 Apr;47(2):301-9. doi: 10.1016/j.ocl.2015.09.005. PMID 26772938
- [Background] Wu JP, Kirk TB, Zheng MH. Study of the collagen structure in the superficial zone and physiological state of articular cartilage using a 3D confocal imaging technique. J Orthop Surg Res. 2008 Jul 17;3:29. doi: 10.1186/1749-799X-3-29. PMID 18637164
- [Background] Xia B, Di Chen, Zhang J, Hu S, Jin H, Tong P. Osteoarthritis pathogenesis: a review of molecular mechanisms. Calcif Tissue Int. 2014 Dec;95(6):495-505. doi: 10.1007/s00223-014-9917-9. Epub 2014 Oct 14. PMID 25311420
- [Background] Zampieri S, Mosole S, Lofler S, Fruhmann H, Burggraf S, Cvecka J, Hamar D, Sedliak M, Tirptakova V, Sarabon N, Mayr W, Kern H. Physical Exercise in Aging: Nine Weeks of Leg Press or Electrical Stimulation Training in 70 Years Old Sedentary Elderly People. Eur J Transl Myol. 2015 Aug 25;25(4):237-42. doi: 10.4081/ejtm.2015.5374. eCollection 2015 Aug 24. PMID 26913162
- [Background] Zeng C, Li H, Yang T, Deng ZH, Yang Y, Zhang Y, Lei GH. Electrical stimulation for pain relief in knee osteoarthritis: systematic review and network meta-analysis. Osteoarthritis Cartilage. 2015 Feb;23(2):189-202. doi: 10.1016/j.joca.2014.11.014. Epub 2014 Nov 26. PMID 25497083
- [Background] Lun V, Marsh A, Bray R, Lindsay D, Wiley P. Efficacy of Hip Strengthening Exercises Compared With Leg Strengthening Exercises on Knee Pain, Function, and Quality of Life in Patients With Knee Osteoarthritis. Clin J Sport Med. 2015 Nov;25(6):509-17. doi: 10.1097/JSM.0000000000000170. PMID 25591130